CLINICAL TRIAL: NCT06913426
Title: Effects of Pelvic Tilt Exercises Along With Hip and Knee Focused Exercises on Patients With Patellofemoral Pain Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/797
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Papaverine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Tilt, Hip and Knee Focused Exercises (Intervention Group) (Experimental)
  Interventions: Combination Product: Pelvic Tilt, Hip and Knee Focused Exercises (Intervention Group)
- Hip and Knee Focused Exercises(Control Group) (Active Comparator)
  Interventions: Diagnostic Test: Hip and Knee Focused Exercises(Control Group)

INTERVENTIONS:
Combination Product: Pelvic Tilt, Hip and Knee Focused Exercises (Intervention Group) — The treatment program is between one to six weeks with strictly 18 sessions with at least thrice in a week to give room to recuperate from muscle fatigue. This protocol is set in a 45 minutes session that involves a series of exercises and stretches. The quadriceps muscles strengthening exercises, hamstring and the calf raising workouts such as the hamstring curls and heel raise are done in 3 sets of 10-15 reps. Patellofemoral joint mobilization which should not last more than 2-3 minutes due to possible patient discomfort is performed and its primary goal is increasing joint mobility. After that the patient is to perform exercises for pelvic tilt in three approaches, each made in 10 to 15 repetitions.
  Arms: Pelvic Tilt, Hip and Knee Focused Exercises (Intervention Group)
Diagnostic Test: Hip and Knee Focused Exercises(Control Group) — The treatment program covers a time frame of one to six weeks, three sessions a week, total of 18 sessions, over six weeks. Each session takes 45 minutes and contains a schedule of activities. The quadriceps muscles strengthening exercises, hamstring and the calf raising workouts such as the hamstring curls and heel raise are done in 3 sets of 10-15 reps. Patellofemoral joint mobilization which should not last more than 2-3 minutes due to possible patient discomfort is performed and its primary goal is increasing joint mobility. Then Patient performs hip exercises; hip abductor as well as hip extension, which are done in three sets of 10 to 15 repetitions each. Likewise, the knee-focused workouts such as quad sets, straight leg raises and step-up are conducted in the same 3 sets of 10-15 repetitions style. Static flexibility exercises includes Hip Flexor Stretch, IT Band Stretch and these exercises are performed with 5 sets of 30 seconds.
  Arms: Hip and Knee Focused Exercises(Control Group)

SUMMARY:
This study is designed as a Randomized Controlled Trial to be conducted at the CRC Department of Chaudhary Muhammad Akram Teaching and research Hospital, Lahore.

DETAILED DESCRIPTION:
A total of 48 participants will be recruited accounting for a 10% dropout rate (42+6=48) and equally divided into two groups 24 participants in each group: Group A(Intervention) and Group B(Control). Participants will be selected based on inclusion criteria which includes individuals aged 35-55 years with a clinical diagnosis of Patellofemoral Pain Syndrome (positive Patellar Compression Test) symptoms persisting for at least 6 weeks to 6 months and moderate-to-severe knee pain (NPRS ≥ 4). They must also be willing to comply with study protocols. Exclusion criteria include recent knee surgery, other knee conditions (e.g., ligament injuries or severe osteoarthritis), and neurological disorders affecting movement or cognition.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a clinical diagnosis of Patellofemoral Pain Syndrome.
* Participants should be aged between 35 and 55 years, as this is the typical age group affected by PFPS and will help standardize the sample.
* Individuals with a BMI ranging from 18 to 25 kg/m2.
* Participants should have had symptoms of PFPS for at least 6 weeks to 6 months, ensuring the condition is subacute and chronic.
* Knee Pain Severity: Patients must report moderate to severe knee pain (e.g., pain score ≥ 4 on a 0-10 pain scale) to assess the effectiveness of rehabilitation interventions.
* Participants must be willing to engage in the prescribed exercise program and comply with study protocols including follow-up assessments.

Exclusion Criteria:

* Individuals who have undergone knee surgery within the last 6 months, as post-surgical rehabilitation could interfere with the study outcomes and confound results. Patients with other knee conditions, such as ligament injuries (e.g., ACL or MCL tears), meniscal tears or osteoarthritis, which could significantly affect rehabilitation or complicate the assessment of PFPS.
* Individuals with severe knee osteoarthritis (e.g., Kellgren-Lawrence grade 3 or 4) as it may impact the treatment response and differ from the typical PFPS rehabilitation approach.
* Individuals with neurological conditions (e.g., stroke, multiple sclerosis or peripheral neuropathy) that affect movement, balance or cognition making participation in rehabilitation exercises unsafe or difficult.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Patellar Grind Test | 12 Months
  The Patellar Grind Test, also known as Clarke's Sign, is a physical examination used to assess patellofemoral joint pain, involving compression of the patella while the patient contracts their quadriceps, with a positive test indicated by pain or grinding
Numeric Pain Rating Scale (NPRS) | 12 Months
  Knee Pain during Daily Activities and Exercises is assessed using the numeric pain rating scale for Pain. It is highly reliable based on construct validity and it really measures the degrees of pain and possess significant test-retest reliability.
  The lowest value, 0, means that the patient felt no pain at all. The highest value 10, means the worse pain that could be conceived.
Kujala Patellofemoral Score (Anterior Knee Pain Scale) | 12 Months
  Kujala Patellofemoral Score better known as Anterior Knee Pain Scale is self-administered questioner aimed at quantifying the severity of AKP and restriction in activity related to PFPS. It has 13 questions which are focused on certain activity or symptom.
  Scoring:
  Each question is scored, and the total ranges from 0 to 100:
  0: Higher severity of the symptoms and higher degree of self-implemented limitations.
  100: No symptoms, normal function. Interpretation of Scores. 85-100: Perfect working, few indications. 70-84: Good function, mild symptoms. 50-69: Sufficient function, phenomena slightly manifesting themselves. Below 50: Low, worst.

CONTACTS AND LOCATIONS:
Locations (1):
- Superior University CRC, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No